CLINICAL TRIAL: NCT06745635
Title: A Multifaceted Intervention on Reducing Immunization Errors: a Pragmatic, Stepped-wedge, Cluster Randomized Trial
Brief Title: A Multifaceted Intervention on Reducing Immunization Errors
Acronym: THEIA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Collaborators: Ministry of Health, Brazil (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: THEIA trial
Record Dates: First submitted 2024-12-11; First posted 2024-12-20 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-12

CONDITIONS: Vaccines; Vaccines Adverse Reaction; Vaccine Practice
Keywords: Cluster-randomized controlled trial; Multifaceted intervention; Quality improvement in immunization; Vaccination errors; Vaccination safety; Primary health care; Vaccination room management; Cold chain management; Public health improvement; Health systems implementation

STUDY DESIGN:
Intervention Model Description: A Stepped-Wedge Cluster Randomized Trial (SW-CRT) is a type of clinical trial in which the intervention is progressively implemented across clusters (groups) over time in a staggered and randomized manner. Initially, all clusters start in the control group, and in successive steps, one or more clusters are randomly selected to receive the intervention. This process continues until all clusters have been exposed to the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Care Group (Other): This arm will continue to follow the routine activities and standard procedures established by the public health system.
  Interventions: Other: Usual Care
- Multifaceted Intervention Group (Other): This group will implement a multifaceted quality improvement and process strategy composed of:
  Video-based training on vaccine management. Development of an optimized Cold Chain Manual, streamlining guidelines for vaccine handling.
  Technical documents providing comprehensive guidance on the appropriate management of vaccines and their respective immunization schedules.
  Technical documents addressing the management of errors identified post-vaccination and offering recommendations for public guidance
  Interventions: Other: Multifaceted intervention

INTERVENTIONS:
Other: Usual Care — Usual care for immunizations.
  Arms: Usual Care Group
Other: Multifaceted intervention — The multifaceted quality improvement intervention includes: video-based training on vaccine management in SUS, an optimized Cold Chain Manual schema, technical documents on proper vaccine handling and immunization schedules, and checklists for managing post-vaccination errors and corrective procedures. Videos will focus on six key points (right person, vaccine, dose, time, route, and documentation), with each lasting about 2 minutes and accessible on-demand. The Cold Chain schema will cover storage, monitoring, transport, conservation, and handling, with checklists for each category. Standardized technical documents will align with video themes, ensuring protocol adherence. An error identification and management schema will address issues like improper vaccine administration, cold chain violations, and incorrect dosages. This schema will be reviewed by staff and made available in health units.
  Arms: Multifaceted Intervention Group

SUMMARY:
The goal of this trial is to reduce the general error related to vaccines and immunizations (composited on secondary endpoint), after 11 moths of folow-up after cluster randomization and stepped wedge on primary care on brazilian public health.

The main questions it aims to answer are:

1. To evaluate the effectiveness of a multifaceted intervention in vaccination rooms in reducing vaccination errors.
2. To describe the rate of adverse events following immunization (AEFI) and the associated factors.

DETAILED DESCRIPTION:
Researchers will compare two times in a Stepped Wedge design:

1. Usual Care :All sites will follow the standard practices for vaccine management and immunization in health units with vaccination rooms during 1 month.

   All sites will be randomized into 11 steps (corresponding to the number of stages required to complete the 12-month study). At each step, 8 clusters (each containing one immunization service within a primary care facility) will receive the intervention."
2. Multifaceted Strategy :*This time will implement a multifaceted quality improvement and process strategy composed of:

   * Video-based training on vaccine management.
   * Development of an optimized Cold Chain Manual, streamlining guidelines for vaccine handling.
   * Technical documents providing comprehensive guidance on the appropriate management of vaccines and their respective immunization schedules.
   * Technical documentsaddressing the management of errors identified post-vaccination and offering recommendations for public guidance.

ELIGIBILITY:
Cluster Inclusion Criteria

* Health units with vaccination rooms administering at least 2,000 doses of vaccines/immunobiologicals per month,

Cluster Exclusion Criteria

* Primary health units that do not provide consistent vaccination services to the population.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-07-03 (Estimated); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Reduction of overall errors attributable to vaccination and immunization processes. | From Randomization to the end of Follow-up (12 months)
  The primary composite outcome is defined as the reduction of overall errors attributable to vaccination and immunization processes, including: dilution errors, administration of vaccines outside the recommended age, errors related to inappropriate intervals between doses/vaccines, errors in the use of immunobiologicals, errors related to repeated doses, administration of vaccines not recommended during pregnancy, errors in the storage and handling of vaccines and immunobiologicals, and administration of vaccines via incorrect routes.

SECONDARY OUTCOMES:
incidence of the components of the primary outcome | Through study completion, an average of 1 year
  Rate of the components of the primary outcome.

OTHER OUTCOMES:
Primary Secondary Outcome - Incidence of reported Adverse Events Following Immunization | From Randomization to the end of Follow-up (12 months)
  Incidence of reported Adverse Events Following Immunization (AEFI) in the studied health units-AEFIs recorded either spontaneously or through active surveillance within the health units during the study period.
Exploratory Objective - Economical impact of strategy for reduce the error of immunization | Through study completion, an average of 1 year
  Cost-Effectiveness - Economical impact of strategy for reduce the error of immunization as basis for public vaccination policy justification -

CONTACTS AND LOCATIONS:
Overall Officials: Henrique A Fonseca, ScD, PhD, Study Chair — Hospital Albert Einstein
Locations (1):
- Hospital Israelita Albert Einstein, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No